CLINICAL TRIAL: NCT06455579
Title: Bedtime Stories: A Sleep Health Education Program for Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Allan & Gill Gray Foundation (Unknown)
Responsible Party: Principal Investigator, Judith Owens, Professor of Neurology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00044533
Record Dates: First submitted 2024-05-22; First posted 2024-06-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sleep; Health-Related Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep Health Education Program for Healthcare Providers (Experimental): The BTS-HP is an online sleep health education program supported by the Boston Children's Hospital Department of Education (CE Courses - BCH Education (childrenshospital.org). The provider will also receive access to an educational webinar on Melatonin. The provider can participate all modules and the webinar in one sitting or overtime.
  Interventions: Behavioral: Bedtime Stories Sleep Health Education Program for community healthcare providers (BTS-HP)

INTERVENTIONS:
Behavioral: Bedtime Stories Sleep Health Education Program for community healthcare providers (BTS-HP) — The sleep health education program includes 6 educational modules on different topics related to sleep health: (1) Basics of Sleep, 2) Sleep and Development, 3) Sleep Health, 4) Consequences of Deficient Sleep, 5) Sleep Health Disparities, and 6) Sleep Screening and Evaluation.

SUMMARY:
This is a pilot intervention of the Bedtime Stories Sleep Health Education Program for healthcare providers serving school aged children and their caregivers. The intervention uses a pre-post design across participants.

DETAILED DESCRIPTION:
To date, there are no established sleep health education programs for healthcare providers. To address this gap, the investigators previously conducted semi-structured interviews with community-based healthcare providers to improve our knowledge and understanding of healthcare providers' attitudes and beliefs about sleep health, factors that may contribute to poor sleep health, and identify potential sleep health promotion strategies for low income, racial and ethnic minority children and their families. Data from those sessions helped to inform and refine content to develop a sleep health education program for community healthcare providers. The purpose of this protocol it assess the effectiveness of the Bedtime Stories Sleep Health Education Program in Community Healthcare Providers (BTS-HP).

Healthcare providers from participating community healthcare centers will be invited to participate. Once a healthcare provider expresses interest in participating, they will receive a REDCap link to provide their informed consent. The provider will then complete a short demographic questionnaire via REDCap. Once the healthcare provider consents and completes the short questionnaire, they will receive a secure link to the Bedtime Stories Sleep Health Education Program for Healthcare Providers (BTS-HP). The BTS-HP is an online sleep health education program supported by the Boston Children's Hospital Department of Education (CE Courses - BCH Education (childrenshospital.org). The provider will also receive access to an educational webinar on Melatonin. The provider can participate all modules and the webinar in one sitting or overtime. Once the provider completes the online modules, they will immediately receive an email with a REDCap link to complete their post-participation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Community Healthcare Provider (physicians, residents, registered nurses, nurse practitioners) at participating community healthcare centers in the Boston area
* Serve families with school-aged (4-10 years of age) children
* English fluency

Exclusion Criteria:

* Community healthcare providers that do not see school-aged children (4-10 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Provider knowledge, perceptions, and practices of sleep health | 1-14 days
  Changes in self-reported knowledge, attitudes, confidence, intent to change practice (questions included in the post participation questionnaire). Retrospective pre-post survey.
  The scale is named "Sleep Questions for Retrospective Pre-Post Survey". The minimum value is 10 and the maximum value is 55. A higher score indicates more confidence in sleep health knowledge (a better outcome).

SECONDARY OUTCOMES:
Provider Acceptability | 1-14 days
  Sample questions BTS-HP experience survey (e.g. questions: How was easy the training to use? How was this training in anticipatory guidance?
Provider Feasibility (number of modules) | 1-14 days
  Monitor access and completion of modules by counting the number of modules accessed and/or completed for each provider through the online portal.
Provider Feasibility (time spent) | 1-14 days
  Monitor access and completion of modules by measuring the time spent on each module for each provider through the online portal.
Provider Feedback on Drafted Content | 1-14 days
  Feedback on their participation and their use of content, sleep health material.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Owens, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owens JA. The practice of pediatric sleep medicine: results of a community survey. Pediatrics. 2001 Sep;108(3):E51. doi: 10.1542/peds.108.3.e51. PMID 11533369
- [Background] Owens JA, Jones C. Parental knowledge of healthy sleep in young children: results of a primary care clinic survey. J Dev Behav Pediatr. 2011 Jul-Aug;32(6):447-53. doi: 10.1097/DBP.0b013e31821bd20b. PMID 21546852
- [Background] Meltzer LJ, Mindell JA. Systematic review and meta-analysis of behavioral interventions for pediatric insomnia. J Pediatr Psychol. 2014 Sep;39(8):932-48. doi: 10.1093/jpepsy/jsu041. Epub 2014 Jun 19. PMID 24947271